CLINICAL TRIAL: NCT03132909
Title: Attitudes and Feelings of Doctors Caring for Their Colleagues: a Qualitative Study in Picardy
Acronym: ATTRESMED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-43 Dr Deschasse
Record Dates: First submitted 2017-04-13; First posted 2017-04-28 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Feelings; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Feelings Determination — Determine the feelings of doctors caring for their colleagues

SUMMARY:
The sick doctor is a patient apart. His right of prescription and his knowledge of semiology easily lead him to self-medication.

DETAILED DESCRIPTION:
The sick doctor is a patient apart. His right of prescription and his knowledge of semiology easily lead him to self-medication. Several factors linked to his profession may also lead to a delay in care: overworking with schedules that are not compatible to organize follow-up, poor access to prevention or occupational medicine for liberal doctors but also modesty And ashamed of being sick (and especially unfit to heal). Specialized centers and specific training courses concerning burnout, addictions and psychiatric pathologies of doctors are currently emerging.

To look after a colleague also seems to imply certain specificities like the sharing of knowledge or the medical vocabulary. The physician-patient relationship may seem easier, but it can also lead to confusion of roles and create ambiguity. In this case, the doctor may feel too close to the doctor-patient to maintain his objectivity and to treat him properly. In the same way, the relationship of trust can be altered by sharing medical knowledge, communication techniques or confidence building which can thus lose their effectiveness.

This physician-caregiver relationship has already been the subject of some qualitative research demonstrating the difficulty from the point of view of the treated. The feelings and attitudes of the doctor caring for his colleague remains a field very little studied. The research hypothesis is that there are specificities to this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Practicing general practitioners, registered with the Order, caring for or having treated other doctors whatever their specialties

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Doctors caring for their colleagues
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Analyze the feelings of doctors who care for their colleagues through a questionnaire | 10 months
  Analyze the feelings of doctors who care for their colleagues through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No